CLINICAL TRIAL: NCT06725888
Title: A Prospective, Multicentre, Open-label, Study to Assess Performance and Safety of the Medical Device Vagitab - T in Rebalancing the Altered Vaginal Flora as Adjuvant Therapy in Patients With Bacterial Vaginosis and in Reducing Incidence of Recurrence During a 3-months Period of Follow-up.
Brief Title: Evaluation of the Medical Device Vagitab - T as Adjuvant Therapy in Patients With Bacterial Vaginosis.
Acronym: Vagitab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: S.I.I.T. Srl (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIIT/VAG/0222
Record Dates: First submitted 2024-11-20; First posted 2024-12-10 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Bacterial Vaginosis (BV); Recurrent Bacterial Vaginosis
Keywords: Bacterial Vaginosis; Recurrent Bacterial Vaginosis; Vaginal microflora; Lactobacillus
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vagitab-T plus metronidazole (the standard treatment for bacterial vaginosis). (Experimental): Vagitab-T for 3 monthly cycles In addition, metronidazole (the standard treatment for bacterial vaginosis) will be administered for seven days.
  Vagitab -T: 1.1 g vaginal tablets; medical device class IIa, already CE marked. The product contains the following components:
  tyndallized probiotic L. plantarum HA-119, lactic acid, and xylo-oligosaccharides, lauryl glucoside, and macrogol 3350
  Metronidazole It is the treatment indicated for Bacterial Vaginosis by the 2021 CDC's Sexually Transmitted Infections Treatment Guidelines.
  Metronidazole will be administered vaginally (as 500 mg vaginal ovules) or orally (as 500 mg tablets)
  Interventions: Device: Vagitab -T vaginal tablets. Components: tyndallized probiotic L. plantarum HA-119, lactic acid, and xylo-oligosaccharides, lauryl glucoside, and macrogol 3350:

INTERVENTIONS:
Device: Vagitab -T vaginal tablets. Components: tyndallized probiotic L. plantarum HA-119, lactic acid, and xylo-oligosaccharides, lauryl glucoside, and macrogol 3350: — Vagitab -T will be used for 3 monthly cycles of 10 days each. Metronidazole will be used for 1 cycle of 7 days at the start of the study
  Metronidazole will be administered as follows:
  500 mg intravaginally once per day for 7 days or 500 mg orally 2 times/day for 7 days

SUMMARY:
This clinical trial is looking at how well and safely the vaginal administration of Vagitab-T works . Vagitab-T is already on the market in several countries in Europe as a medical device.

The main goals of this trial are to see if the recurrence rate of bacterial vaginosis goes down during the study, if it helps balance the altered vaginal flora during antibiotic treatment, if it improves vaginal secretions, and if vaginal microflora return to normal. We'll also ask the participants about their quality of life and whether they think the treatment is safe.

All 30 women will get the same treatment, and there's no comparison group. They'll be treated with Vagitab-T vaginal tablets for three monthly cycles. Also, metronidazole will be taken at the start of the study for seven days.

Participants will sign an informed written consent and we'll visit them at the start (day 0) and end (day 90) of the study. In addition, we'll call them during each of the three cycles of treatment.

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) affects 20-25% of the general population and is the most common cause of vaginal discharge. It is a polymicrobial disease that typically manifests when the protective antibacterial activity of vaginal lactobacilli is impaired, allowing for the overgrowth of anaerobic bacteria and other pathogens, including Gardnerella vaginalis and Mycoplasma hominis. The term "recurrent bacterial vaginosis" (RBV) is used to describe a condition characterized by two to three episodes of bacterial vaginosis (BV) per year. The recurrence rates are as high as 35% within one month, 50% within three months, and 70% within 12 months.

Given the multiplicity of potential risk factors, the aetiology and pathogenesis of BV remain incompletely understood, and the efficacy of current treatment regimens is variable, resulting in high recurrence rates.

A review of the medical literature reveals that no recommended gold-standard therapies have been established, and that the treatments are not always effective, resulting in high recurrence rates. Consequently, the objective of clinical research is to identify safe and effective products that do not disrupt the delicate equilibrium of the vaginal microbiota. It is imperative to commence treatment promptly following antibiotic therapy to impede the formation of a vaginal biofilm.

Recent published reviews and meta-analyses have demonstrated the efficacy of probiotic preparations in the treatment and prevention of BV. These studies suggest that the amount of exogenously applied Lactobacilli may influence the effectiveness of the treatment. The rationale for testing Vagitab-T as an adjuvant product in the treatment of BV and in preventing the recurrences, and consequently in reducing the use of antibiotics without causing resistance, is based primarily on the synergistic association of functional ingredients and mechanism of action. Vagitab-T is a topical intravaginal tablet formulation that employs several components, including tyndallized probiotic L. plantarum HA-119, lactic acid, and xylo-oligosaccharides, lauryl glucoside, and macrogol 3350, employed for the prevention and treatment of vaginal infections of bacterial or mycotic origin, for the facilitation of the regrowth of a healthy microflora, and for the reduction of the symptoms of vaginal dryness. Vagitab-T is classified as a medical device due to the mechanisms of action, which do not involve the use of biocidal, immunostimulant, or pharmacological effects. Additionally, these mechanisms do not interfere with the functions of host cells.

This open, non-randomized trial will be conducted at two clinical sites in Romania. The objective is to evaluate the efficacy, safety, and tolerability of Vagitab-T vaginal tablets in women diagnosed with bacterial vaginosis (BV) according to the Amsel criteria and with a history of recurrent BV (RBV), defined as at least two episodes per year. The patients will be treated with Vagitab-T vaginal tablets for three monthly cycles of 10 days each, with concurrent administration of metronidazole for seven days. The study duration for each patient is 90 days. The sample size has been determined to be 30 evaluable patients, and the investigators intend to screen 33 patients to achieve this number (allowing for three screening failures). The main objectives of the study will be the evaluation of the reduction of recurrence rate of Bacterial Vaginosis during a 3-month cycle treatment, the adjuvant activity in rebalancing the altered vaginal flora during the antibiotic treatment period, and in improving the fluidity of vaginal secretions. Additional objectives will be the evaluation of the rate of return to normality of vaginal microflora, the quality of life, and the safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged from 18 to 65 years (inclusive).
* Patients affected at enrolment by BV diagnosed according to Amsel criteria, candidate to start an antibiotic therapy with metronidazole.
* Patient with a medical history of RBV (at least 2 episodes of BV in the last 12 months including the current episode).
* Patients who are, in the opinion of the Investigator, able to understand the study, cooperate with the study procedures and attend all the study visits.
* Patients who have given their written informed consent to participate in the study.

Exclusion Criteria:

* Patient with a medical history of HIV or any other immunodeficiency.
* Patients working as sex workers.
* Patients with known allergies or intolerance / hypersensitivity to the tested medical device and its components.
* Patients with concomitant menstrual bleeding at baseline.
* Time between the last day of last menses and treatment with metronidazole ≤ 3 days.
* Pregnant, lactating, and lactating amenorrhoeic patients and patients of childbearing potential who are planning a pregnancy or unwilling to use appropriate methods of contraception during the study
* Concomitant use of vaginal tampons.
* Concomitant administration of etonogestrel/ethinyl estradiol vaginal rings or of intrauterine devices.
* Concomitant use of oral or vaginal antibiotic therapy (apart from metronidazole) or any other vaginal therapies or treatment (such as douching, spermicide).
* Concomitant use of oral or vaginal probiotics.
* Patients with any other medical condition that, in the opinion of the Investigator, would compromise participation or be likely to lead to hospitalization during the study.
* Concomitant or previous (in the previous 30 days) participation in any other interventional clinical trials

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female will be included in the study
Enrollment: 30 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-09-23 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Bacterial Vaginosis (BV) Recurrence | 90 days
  BV recurrences will be clinically diagnosed according to the Amsel criteria, which define the presence of BV based on the presence of at least 3 of the following 4 criteria: vaginal pH > 4.5, clue cells on saline wet mount, release of a fishy amine odor when 10% potassium hydroxide is added to a drop of vaginal discharge ("whiff test"), and/or characteristic thin, homogeneous vaginal discharge. The number of BV recurrences in the enrolled population during the 3 months of the study will be compared to the average untreated recurrence rate reported in the medical literature (approximately 50% within 3 months).

SECONDARY OUTCOMES:
Fluidity of vaginal secretion | 90 days
  The subjective rating of vaginal secretion fluidity is determined by patients using a Visual Analog Scale (VAS). The VAS is a horizontal line, 100 mm in length. The left end of the line is marked "0," indicating minimum fluidity, while the right end is marked "100," indicating maximum fluidity. Patients are instructed to mark the point on the line that best represents the fluidity of their secretions. The VAS score is determined by measuring millimeters from the left end of the line to the point marked by the patient. Change is assessed from baseline to 90 days (end of study).
Normality of vaginal flora | 90 days
  It is evaluated by the investigators using the Nugent score. The vaginal smears are plated on a microscope slide in oil immersion and at least 10 high power fields are examined for three bacterial morphotypes: Lactobacillus, Gardnerella, and curved gram rods. Each of these three categories is given a score based on the number of bacteria counted. These three scores are then added together to give a total score from 0 - 10. The score is as follows: 0-3: negative for BV, 4-6: intermediate, and 7+: positive for BV. Samples analysis is performed in a central laboratory.
  Change will be assessed from baseline to 90 days (end of study).
Vaginal Lactobacillus Microbiota | 90 days
  Mucus and cell samples collected from the endocervix by swabbing will be evaluated by optical microscopy using the following classification: normal (numerous pleomorphic lactobacilli, no other bacteria or clue cells or hyphae); partially impaired (population of lactobacilli severely reduced); pathological (lactobacilli severely reduced or absent due to overgrowth of other bacteria or clue cells (>20%) or hyphae).
  Change evaluated from baseline to 90 days (end of study)
Vaginal Discharge | 90 days
  It is evaluated over the past 24 hours using the following 3-point scale: 0 = absent or physiological; 1 = mildly abnormal (abnormal amount with normal color and type); 2 = abnormal amount and abnormal color and type.
Burning | 90 days
  It is rated over the past 24 hours using the following 5-point scale: 0 = not present; 1 = mild; 2 = moderate; 3 = severe; 4 = unbearable
Erythema | 90 days
  It is rated on the following 5-point scale: 0 = no symptoms; 1 = mild; 2 = moderate; 3 = severe: 4 = very severe.
Dyspareunia | 90 days
  It is evaluated using the following dichotomic scale: 0 = absent; 1 = present.
Quality of Life (QoL) | 90 days
  Quality of Life (QoL) is assessed using the SF-12 questionnaire, comprising twelve questions pertaining to the individual's physical and mental health. Each question is scored from 1 to 5, with the total score ranging from 0 to 100. Higher scores indicate better health functioning.
Investigator Overall Performance | 90 days
  It is evaluated using the Investigator Global Assessment of Performance Questionnaire (IGAP). The questionnaire evaluates treatment performance using the following 4-point scale: 1 = very good performance; 2 = good performance; 3 = fair performance; 4 = poor performance.
Patient Overall Performance | 90 days
  It is assessed by the Patient Global Assessment of Performance Questionnaire (PGAP). The questionnaire, evaluates treatment performance using the following 4-point scale 1 = very good performance; 2 = good performance; 3 = fair performance; 4 = poor performance
Investigator Overall Safety | 90 days
  The assessment is conducted using the Investigator Global Assessment of Safety Questionnaire (IGAS). The questionnaire assesses the safety of the treatment in question using a 4-point scale: 1 = very good safety; 2 = good safety; 3 = fair safety; 4 = poor safety.
Patient Overall Safety | 90 days
  The assessment is conducted using the Patient Global Assessment of Safety Questionnaire (PGAS). The questionnaire evaluates the safety of the treatment in question using a 4-point scale: 1 = Excellent safety; 2 = Good safety; 3 = Fair safety; 4 = Poor safety.
Serious Adverse Device Effects / Serious Adverse Events /Adverse Device Effects/ Adverse Events | 90 days
  The number of participants with treatment-related adverse events will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) v 6.0

CONTACTS AND LOCATIONS:
Overall Officials: Attila Fogarassy, MD, Principal Investigator — Gyniclinique - Strada Johann Wolfgang von Goethe nr. 2 - Timisoara (Romania)
Locations (1):
- Gyniclinique - Strada Johann Wolfgang von Goethe nr. 2, Timișoara, Timiș County, Romania